CLINICAL TRIAL: NCT01329003
Title: DNA-damage Pathways in Workers Exposed to Silica (Caesar Stone)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Elizabeth Fairman, Tel Aviv medical center
Other Study IDs: TASMC-11-YS-620-CTIL
Record Dates: First submitted 2011-02-06; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-03

CONDITIONS: Silicosis
Keywords: Silicosis
MeSH Terms: conditions — Silicosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood 20 ml(cc)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- exposed workers: At least six months of occupational exposure to Caesar stone

SUMMARY:
Silicosis is well-known occupational disease caused by free crystalline silica (silicon dioxide) and is marked by inflammation and pulmonary fibrosis. There are cumulative evidences that exposure to Caesar stone (quartz surface products that manufactured from up to 93% quartz, polymer resins and pigments) is particularly dangerous to exposed workers.

Goals: To examine correlation between disease and exposure to Caesar stone and genetic differences regarding genes involved in oxidative stress to understand Genetic susceptibility

DETAILED DESCRIPTION:
It is a sub-study of "DNA-damage biomarkers to monitor and early detect health impairment in workers exposed to Silica (Caesar Stone)" study. Study participants would be recruited during two years of the study. They will be asked to come to a single visit at Pulmonary Laboratory of Tel Aviv Medical Center. During the meeting, participants will be given a precise explanation about the tests they will perform and after signing the informed consent will perform following tests:

1. Induced sputum (IS)
2. Exhaled Breath Condensate
3. Pulmonary function tests (PFTs)
4. Participants will be asked to complete occupational questionnaire

Genetic studies (DNA) will be done from peripheral blood samples (20 ml) to study differences in Heme oxygenase 1 (HO-1) gene sequencing between participants with evidences of clinically definite silicosis according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines and participants without evidences of clinically definite silicosis.DNA samples will be obtained and coded in the same day of a participant visit and after collecting reasonable amount of samples examination of genes of interest will be done.Analysis of data will be done after the completion of data collection and laboratory tests.

Each sample will be given specific code to protect confidentiality of participants. Blood samples, test results and the code key will be kept in different places and only few research staff will have the accessibility to genetic information. In any case employers or any other persons that not included in research staff will not have any accessibility to this information. In this study genetic analysis is not connected to gender, nationality or any other social feature.

ELIGIBILITY:
Inclusion Criteria:

1. male
2. 18-70 years old
3. At least six months of professional exposure to Caesar stone

Exclusion Criteria:

1. Other occupational exposure (welding of any kind)
2. Chronic Obstructive Pulmonary Disease (COPD), tuberculosis, asthma, autoimmune disease in healthy exposed workers
3. Interstitial lung disease in exposed workers with clinically approved silicosis

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least six months of occupational exposure to Caesar stone
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite silicosis according to American Thoracic Society/European Respiratory Society (ATS/ERS)guidelines | one day
  1. Occupational physician examination
  2. Pulmonary function tests (PFTs): The measurement will be performed using standard protocols according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines. Including Lung diffusion testing
  3. Computed Tomography (CT) test if need

SECONDARY OUTCOMES:
Differences in Heme oxygenase 1 (HO-1) gene sequencing | one day
  Genetic studies (DNA) will be done from peripheral blood samples (20 ml) to study differences in Heme oxygenase 1 (HO-1) gene sequencing between participants with evidences of clinically definite silicosis according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines and participants without evidences of clinically definite silicosis

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Shwartz, MD, Principal Investigator — Tel Aviv medical center. Pulmonary and Allergy department
Locations (1):
- Pulmonary Laboratory of Tel Aviv Sourasky Medical Center, Tel Aviv, Israel